CLINICAL TRIAL: NCT06956495
Title: Efficacy and Tolerability of Tasipimidine After 3 Repeated Bed-Time Doses in Patients With Insomnia Disorder With a 4-week Extension Part
Brief Title: Efficacy and Tolerability of Tasipimidine in Sleepless Patients
Acronym: Unitas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 3110012; 2022-502483-21-00 (EU CTIS Number); ISRCTN35042256 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Part 1: escalating dose levels administered to sequential cohorts of subjects. Part 2: participants randomised to parallel groups receiving one of the selected dose levels or placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tasipimidine Dose level 1 (Experimental): Dose level 1
  Interventions: Drug: Tasipimidine
- Tasipimidine Dose level 2 (Experimental): Dose level 2
  Interventions: Drug: Tasipimidine
- Tasipimidine Dose level 3 (Experimental): Dose level 3
  Interventions: Drug: Tasipimidine
- Placebo (Placebo Comparator): Tasipimidine Placebo
  Interventions: Drug: Tasipimidine placebo
- Tasipimidine Dose level 4 (Experimental): Dose level 4
  Interventions: Drug: Tasipimidine

INTERVENTIONS:
Drug: Tasipimidine — Tasipimidine solution
  Other Names: ODM-105
  Arms: Tasipimidine Dose level 1; Tasipimidine Dose level 2; Tasipimidine Dose level 3; Tasipimidine Dose level 4
Drug: Tasipimidine placebo — Tasipimidine placebo solution
  Other Names: ODM-105 placebo
  Arms: Placebo

SUMMARY:
The goal of this trial is to learn if tasipimidine will help in the treatment of insomnia and how safe it is to use in sleepless people. Researchers will compare tasipimidine to a placebo (a look-alike substance that contains no drug) to see if tasipimidine works to treat insomnia. The trial consists of 2 consecutive parts and participants will be included either in Part 1 or Part 2. Part 2 will start only after Part 1 completion. Both parts include a screening period (up to 6 weeks), a treatment period (3 consecutive days and nights) and a post-treatment period (up to 10 days). Part 2 includes an additional 4 week extension part, where the participants take tasipimidine or placebo every evening at home and return to the sleep clinic for 2 last treatment nights. Participants will use equipment to record sleep parameters both at sleep clinic and home (Part 2) and a sleep diary is used.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (IC) for participation in the study.
* Male or female subjects with age between 18 and 65 years.
* Insomnia disorder
* Self-reported history of the following on at least 3 nights per week and for at least 3 months prior to the screening: ≥ 30 minutes to fall asleep, subjective total sleep time ≤ 6 hours.
* Insomnia Severity Index© (ISI©) score ≥ 15 in Part 1 and ≥ 11 in Part 2.
* Usual bedtime between 21:00 and 02:00.
* Regular time in bed between 6 and 9 hours.
* Meeting predefined sleep parameter criteria in sleep recording on the 2 screening nights.
* Highly effective contraception.

Exclusion Criteria:

* Body mass index below 18.5 or above 40.0 kg/m2.
* Daytime napping ≥ 1 hour per day, and ≥ 3 days per week.
* Shift work within 2 weeks prior to the screening visit, or planned shift work during the study.
* Travel across ≥ 3 time zones within 2 weeks prior to the screening visit, or planned travel across ≥ 3 time zones during the study.
* Use of certain medications affecting central nervous system, e.g. sedatives or stimulans.
* Start of other new chronic medication within 14 days prior screening nights and planned change to an ongoing chronic medication during the study.
* Cognitive behavioural therapy (CBT) is allowed if the CBT started at least 1 month prior to the 1st screening night and the subject agreed to continue the CBT throughout the study.
* Diagnosed sleep-related breathing disorder, including chronic obstructive pulmonary disease and sleep apnoea.
* Acute or unstable psychiatric conditions.
* Alcohol or substance use disorder within 2 years prior to the screening visit or inability to refrain from drinking alcohol for at least 3 consecutive days.
* Significant cardiac disease.
* Significant postural hypotension.
* Heavy tobacco or other nicotine containing product use.
* Caffeine consumption ≥ 600 mg per day or regular caffeine consumption after 4 p.m.
* Heart rate < 50 bpm or > 100 bpm.
* Systolic blood pressure < 100 or > 160 mmHg or diastolic blood pressure < 50 or > 100 mmHg
* Abnormal 12-lead ECG finding.
* Significant abnormal laboratory findings including positive drug screen and presence of alcohol in breath test.
* Pre-planned elective surgery.
* Pregnant or lactating females.
* Blood donation or loss of significant amount of blood prior to the study.
* Participation in a drug study within 60 days prior to the study.
* Restless legs syndrome, circadian rhythm disorder, REM behaviour disorder, or narcolepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Wake after sleep onset (WASO) combined from Part 1 and Part 2 | Treatment Day 1 and 2
  Assessed with polysomnography (PSG) for Day 1 and Day 2 data combined from Part 1 and Part 2
Latency to persistent sleep (LPS) combined from Part 1 and Part 2 | Treatment Day 1 and 2
  Assessed with polysomnography (PSG) for Day 1 and Day 2 data combined from Part 1 and Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Terveystalo Helsinki Uniklinikka, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No